CLINICAL TRIAL: NCT05990829
Title: Compare the Efficacy of VItrectomy Combined With DExamethasone Implant Versus With Aflibercept in DME Patients Diagnosed by Intraoperative OCT (the VIDEO Study): Study Protocol for a Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Eye Hospital (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Bojie Hu, Professor, Tianjin Medical University Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TianjinMUEHhbj001
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2023-08

CONDITIONS: Diabetic Macular Edema; Pars Plana Vitrectomy; Dexamethasone Intravitreal Implant; Intraoperative Optical Coherence Tomography
MeSH Terms: interventions — Calcium Dobesilate; aflibercept

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozurdex group (Experimental): Standard 25-gauge pars plana vitrectomy (PPV) will be performed under retrobulbar anaesthesia using high-speed vitrectomy system. Clear all the vitreous hemorrhage and proliferative membrane during PPV operation, panretinal photocoagulation should be completed. The vitreous cavity will be filled with balanced salt solution. An injection of Ozurdex will be performed at the end of the surgery.
  Interventions: Drug: Ozurdex
- Aflibercept group (Active Comparator): Standard 25-gauge pars plana vitrectomy (PPV) will be performed under retrobulbar anaesthesia using high-speed vitrectomy system. Clear all the vitreous hemorrhage and proliferative membrane during PPV operation, panretinal photocoagulation should be completed. The vitreous cavity will be filled with balanced salt solution. An injection of aflibercept will be performed at the end of the surgery.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Ozurdex — Standard 25-gauge pars plana vitrectomy (PPV) will be performed under retrobulbar anaesthesia using high-speed vitrectomy system. Clear all the vitreous hemorrhage and proliferative membrane during PPV operation, panretinal photocoagulation (PRP) should be completed. The vitreous cavity will be filled with balanced salt solution. An injection of Ozurdex will be performed at the end of the surgery.
  Arms: Ozurdex group
Drug: Aflibercept — Standard 25-gauge pars plana vitrectomy (PPV) will be performed under retrobulbar anaesthesia using high-speed vitrectomy system. Clear all the vitreous hemorrhage and proliferative membrane during PPV operation, panretinal photocoagulation (PRP) should be completed. The vitreous cavity will be filled with balanced salt solution. An injection of aflibercept will be performed at the end of the surgery.
  Arms: Aflibercept group

SUMMARY:
Diabetic macular edema (DME) is the main cause of severe vision loss in diabetic retinopathy. Intravitreal injection of anti-vascular endothelial growth factor (VEGF) and Ozurdex are two safe and effective ways to treat DME. Pars plana vitrectomy is mainly suitable for the treatment of unabsorbed vitreous hemorrhage (VH) and tractional retinal detachment caused by proliferative diabetic retinopathy (PDR). Intraoperative optical coherence tomography (OCT), a diagnostic device, can be used to evaluate the potential condition of the retina. Many patients with PDR have unclear refractive stroma due to VH and other reasons, so preoperative OCT cannot give a clear diagnosis, so the use of intraoperative OCT can judge whether the patients are complicated with DME and give corresponding treatment. The purpose of this study is to explore the prognosis of patients with DME diagnosed by OCT during PPV and treated with PPV combined with aflibercept or PPV combined with Ozurdex, and to observe and compare the postoperative anatomical results, functional results, times of reinjections and the occurrence of adverse events between the two groups, in order to provide accurate treatment for patients, reduce the frequency of postoperative vitreous injection and lighten the burden of patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age;
* Patients and their families fully understand the research and must sign an informed consent form;
* Patients have a history of diabetes and were diagnosed with PDR by ophthalmic examination;
* Haemoglobin A1c (HbA1c) levels of <10% within 3 months;
* No contraindication of vitrectomy;
* Pseudophakia or this operation is combined with phacoemulsification and lens implantation;
* Diagnosed with DME by intraoperative optical coherence tomography during vitrectomy

Exclusion Criteria:

* The follow-up period is less than 6 months;
* Patients need gas or silicon oil tamponade;
* Patients with rubeosis iridis, neovascular glaucoma and endophthalmitis;
* Patients with other intraocular surgeries (except cataract surgery with no ruptured posterior lens capsule);
* Patients with other retinal diseases (i.e., age-related macular degeneration, retinal vein occlusion);
* Patients received intravitreal Ozurdex three months prior to screening or anti-VEGF injection one month prior to screening;
* Patients with uncontrolled systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Average change in central foveal thickness (CFT) | 1, 3, 6 month postoperatively
  Three-dimensional swept source optical coherence tomography (SS-OCT)

SECONDARY OUTCOMES:
Average change in best corrected visual acuity (BCVA) | 1, 3, 6 month postoperatively
  Early Treatment Diabetic Retinopathy Study (ETDRS) Alphabet Chart
Number of reinjections | 6 months postoperatively
  Each participant will receive pro re nata therapy, with regular monitoring for 6 months, at least 3 months apart for the study group and 1 month apart for the control group. Further treatment will be performed if the following criteria are met: (1) existence of recent or persisting cystoid retinal lesions; (2) a decrease of no less than 5 Early Treatment Diabetic Retinopathy Study (ETDRS) letters in BCVA; and (3) an increase of 50 m or more in central foveal thickness (CFT) compared with the best value previously achieved.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin medical university eye hosipital, Tianjin, Tianjin Municipality, China